CLINICAL TRIAL: NCT05529498
Title: Effect of High Intensity Interval Gait Training on Ambulation in MS
Brief Title: High Intensity Interval Gait Training in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: City University of New York (Other)
Responsible Party: Principal Investigator, Herbert Karpatkin, Associate Professor, City University of New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CityUNewYork
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis,Gait, Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 2 group pretest postest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): High intensity interval gait training
  Interventions: Behavioral: High Intensity Interval gait training
- Control (Active Comparator): Moderate intesnity continuous gait training
  Interventions: Behavioral: Moderate paced continuous gait training

INTERVENTIONS:
Behavioral: Moderate paced continuous gait training — walking continuously for 20 minutes at a moderate pace
  Arms: Control
Behavioral: High Intensity Interval gait training — 20 minutes of interspersing 30 seconds of fast walking with 1 minute of rest
  Arms: Experimental

SUMMARY:
Over 90% of persons with MS (pwMS) complain of difficulty with walking. High intensity interval gait training (HIIGT), where persons alternate brief periods of walking at high speeds with periods of rest has been found to improve walking in other neurologic diagnoses. However its impact on pwMS is not known. Most gait training in MS is done continuously at a slower pace. The purpose of this study is to compare the effects of HIIGT to traditional Moderate Intensity Continuous Gait Training (MICGT) in pwMS.

DETAILED DESCRIPTION:
Purpose: To determine whether pwMS will have greater improvements in gait with HIIGT as compared to MICGT.

Primary Question: Does HIIGT results in greater improvements in gait parameters in pwMS than MICGT? Secondary question: Will HIIGT result in greater improvements in balance, lower extremity strength, lower extremity range of motion and HR when compared to MICGT in pwMS?

Hypothesis: HIIGT will result in greater improvements in gait parameters in pwMS than MICGT.

Justification: Previous research has shown that MICGT, moderate intensity interval training and high intensity non-gait interval training is effective in pwMS (1)(2). HIIGT has been shown to be effective in persons with stroke (3) but the effects of HIIGT on pwMS are not known.

Outcomes and dissemination of information: We will present our findings at national conferences and submit manuscripts of our findings to the appropriate peer reviewed journal.

The answers to our research questions will be found by using a randomized controlled to group people pretest post test design.

1. - INFORMED CONSENT: Upon entering Hunter College Physical Therapy department, participants will be greeted by dr. Karpatkin and provided with an informed consent form outlining the purpose of the study, the length of the study, the potential risks, and the procedures.
2. - COLLECTION OF DEMOGRAPHICS: Participants will fill out a questionnaire collecting demographics and subject characteristics information, such as age, gender, race, phenotype of MS, ambulatory device used, medications used, years since diagnosis.
3. - COLLECTION OF SELF REPORT MEASURES: Patients will then will out the following self report questionnaires Multiple Sclerosis Impact Scale 29 (MSIS 29): The MSIS 29 is a questionnaire asking for participants' views about the impact of MS on their day-to-day life, measuring coordination, fatigue, flexibility, muscle performance, muscle tone/spasticity, balance/falls, reach and grasp, self-care, health and wellness, leisure, quality of life, role function, social function, work in pwMS.

The Fatigue Severity Scale (FSS): The FSS is a short questionnaire that requires you to rate your level of fatigue. The FSS questionnaire contains nine statements that rate the severity of your fatigue symptoms. Read each statement and circle a number from 1 to 7, based on how accurately it reflects your condition during the past week and the extent to which you agree or disagree that the statement applies to you.

12 Item MS Walking Scale (MSWS-12): is a self-report measure of the impact that MS has on an individual's ambulation. The participants read each statement and report how much MS has limited them in the past two weeks on a scale of 1 to 5.

4 - 6 minute walk test (6MWT): The 6MWT measures the distance an individual is able to walk over a total of six minutes on a leveled surface indoors. The goal is for the individual to walk as far as possible in six minutes. The individual is allowed to self-pace and rest as needed as they traverse back and forth along a marked walkway. We will also be measuring the distance walked in each minute of the test and participants heart rate before, during and after the test.

5 - The Functional Gait Assessment (FGA): is used to assess postural stability and balance during different tasks in populations of pwMS, Parkinson disease, spinal cord injuries, stroke diagnosis, and vestibular disorders. FGA is a modification of the Dynamic Gait Index and was created to help decrease the ceiling effect and improve reliability.

6 - Hand Held Dynamometry (HHD): is used to measure participants' strength in hip flexion, hip extension, knee flexion, knee extension, ankle plantarflexion and dorsiflexion. Measurements will be taken using a dynamometer.

7 - Goniometry: is used to measure ranges of motion for participants' hip flexion, hip extension, knee flexion, knee extension, ankle plantarflexion, and ankle dorsiflexion. Measurements will be taken using a standard goniometer.

8 - RANDOMIZATION INTO HIIGT GROUP AND MICGT GROUP: After collecting the information from the questionnaires, the participants who meet the inclusion criteria will be randomly assigned each participant into either the HIIGT or MICGT group, with each group having an equal number of participants per group. Randomization will be achieved by the participant pulling odd or even numbers out of a hat. An even number will be placed in the HIIGT group and an odd number into the MICGT group. Since the HIIGT represents a novel therapy it will be considered the experimental group. Since the MICGT represents the standard of care it will be considered the control group 7 - DESCRIPTION OF HIIGT PROTOCOL: The protocol for HIIGT will be a total of 4 to 5 weeks including 4 weeks of the intervention, one day of pre-testing and one day of post-testing. Training entails a total of 25 minutes work with 3 minutes warm up of gentle walking, then multiple rounds of 30 seconds of fast walking followed by 60 seconds of seated rest. Fast walking will be defined to the participant as walking the fastest they can comfortably. The participants will complete the cycle of 30 seconds work with 60 seconds rest until they get to 23 minutes of total exercise and then a 2 minute cool down to make 25 minutes of total work. During the intervention each participant's heart rate, Rate of Perceived Exertion, and distance walked will be recorded with a measuring wheel. During the entire protocol, Dr. Karpatkin will be guarding the participant and a wheelchair will be following the participant.

8- DESCRIPTION OF MICGT PROTOCOL: The protocol for MICGT will be a total of 4 to 5 weeks including 4 weeks for the intervention, one day for pre-testing, and one for post-testing. They will engage in continuous moderate walking for 25 minutes per session, 3 times a week for 4 weeks. Moderate walking is defined as a pace the participant is able to comfortably maintain for the 25 minutes. Dr. Karpatkin will be guarding during the full training, and a wheel chair will follow behind the participant. During the intervention each participant's heart rate, Rate of Perceived Exertion, and distance walked will be recorded with a measuring wheel.

9 - POST-TEST PROTOCOL: The post-test protocol will be the same as the pre-test. Each participant will complete the 6MWT, HHD for the lower extremity, Goniometric measures for the lower extremity, and the FGA.

Gate endurance will be operationally defined by performance on the six minute walk test.

Fatigue will also be operationally defined by performance on the six minute walk test.

Balance performance will be operationally defined by performance on the functional gait assessment tool. Lower extremity strength will be operationally defined as performance on handheld dynamometry.

Lower extremity range of motion improvements will be operationally defined as pretest post test improvements in goniometry.

Improvements in heart rate will be measured using pulse oximetry.

Data analysis plan:For all primary outcomes with ratio level data, we will conduct a 2X2 mixed-factor Analysis of Variance (ANOVA). The between-factor will be group type (HIIGT vs MIGGT) and the within-factor will be time (pre-test vs post-test). For the FGA scores (ordinal level data), we will use Generalized Estimating Equations GEEs instead.

We expect a homogenous sample in terms of age, gender, disease severity, and years since onset. However, prior to conducting statistical analyses, we will test the relationship between subject age, disease severity, and years since onset with primary outcome measures using Pearsons correlations (for ratio data) and Spearman's rank correlation (for ordinal data). We will use unpaired t-tests to compare differences in outcome measures between males and females. If any of the subject-characteristic measures have a significant effect on the primary outcome measures, they will be included as covariates or factors in the ANOVA model or GEEs

ELIGIBILITY:
Inclusion Criteria: Persons diagnosed with Multiple Sclerosis. Rationale:because we are studying effects of the intervention on participant with MS

* The ability to walk for 6 minutes continuously with or without assistive device. Rationale:we are using the 6MWT as our primary outcome measure
* The ability to read, understand and sign a consent form so that they are able to understand the study we are doing
* Above the age of 18 because they have to be able to give consent for the study
* English speaking as we do not have the resources for translation for the multiple sessions this study entails

Exclusion Criteria:Any cardiopulmonary, orthopedic, or non-MS neurologic disease as we are only examining the effects of MS and need to rule out the impact of other conditions

* Report of a recent exacerbation. Rationale: the impact of the rationale can interfere with the impact of the independent variables

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | 6 minutes
  Distance covered during continuous walking for 6 minutes

SECONDARY OUTCOMES:
Finctional gait assessment | 10 minutes
  balance during walking

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided